CLINICAL TRIAL: NCT00944125
Title: Dual Site LV Pacing Study: Prospective Randomized Blinded Crossover Study of Patients Meeting Current CRT-D Indication to be Implanted With Dual LV Pacing Leads and Paced Chronically for at Least 6 Months Post-implant.
Brief Title: Dual Site Left Ventricular (LV) Pacing
Acronym: DIVA
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: for administrative reasons (no safety concerns), no analysis completed
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: L-08-166
Record Dates: First submitted 2009-07-17; First posted 2009-07-23 (Estimated); Results first posted 2016-03-21 (Estimated); Last update posted 2024-10-21 (Actual); Status verified 2016-03

CONDITIONS: Congestive Heart Failure; LV Dysfunction
MeSH Terms: conditions — Heart Failure; Ventricular Dysfunction, Left

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual Site LV Pacing (Active Comparator): Prospective randomized blinded crossover study of patients meeting current CRT-D indication implanted with Dual LV pacing leads compared to BiV pacing.
  Interventions: Device: Dual Site LV Pacing; Device: BiV Pacing
- BiV Pacing (Active Comparator): Prospective randomized blinded crossover study of patients meeting current CRT-D indication implanted with Dual LV pacing leads compared to BiV pacing.
  Interventions: Device: Dual Site LV Pacing; Device: BiV Pacing

INTERVENTIONS:
Device: Dual Site LV Pacing — Dual Site LV Pacing vs. BiV Pacing for a total of six months which includes two three crossover periods.
Device: BiV Pacing — Dual Site LV Pacing vs. BiV Pacing for a total of six months which includes two three crossover periods.

SUMMARY:
The purpose of this study is to compare Dual LV (left ventricular) pacing to standard single LV pacing (BiV pacing) to see if Dual LV pacing:

1. Improves the way the heart's left ventricle functions
2. Decreases the number of hospital and clinic visits for heart failure related symptoms
3. Slows the rate patients experience certain heart failure symptoms
4. Reduces uncoordinated heart contractions

ELIGIBILITY:
Inclusion Criteria:

* Moderate or severe heart failure, defined as NYHA Class III-IV despite optimal pharmacological heart failure therapy
* On heart failure medical regimen (beta blockers and ACE-I or ARB's) for at least one month before randomization
* A 12-lead electrocardiogram (ECG) obtained no more than 90 days prior to enrollment documenting a QRS duration > 120 ms
* Left ventricular ejection fraction (LVEF) < 35% or equal
* Willing and capable of undergoing the device implant procedure and participating in all testing associated with this clinical study
* Have a life expectancy of more than 180 days, per physician discretion
* Age 40 or above, ensuring of legal age to give informed consent specific to state and national law

Exclusion Criteria:

* Have had previous cardiac resynchronization therapy or a previous coronary venous lead
* Unable to perform a Six-Minute Hall Walk (6MHW) Test
* Have an atrial tachyarrhythmia that is permanent (i.e., does not terminate spontaneously and cannot be terminated with medical intervention)without CHB or planned AVJ ablation prior to randomization
* Have an atrial tachyarrhythmia that is persistent (i.e. can be terminated with medical intervention, but does not terminate spontaneously) without planned and successful cardioversion prior to randomization (patients with unsuccessful cardioversions and no AVJ Ablation will be exited.)
* Have hypertrophic obstructive cardiomyopathy or infiltrative cardiomyopathy (e.g., amyloidosis, sarcoidosis)
* Have a mechanical tricuspid prosthesis
* Has severe aortic or mitral stenosis
* Enrolled in any concurrent study that may confound the results of this study
* Patients who are or suspect they may be pregnant or plan to become pregnant

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2009-06; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Imran K Niazi, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Aurora Cardiovascular Services, Lake Geneva, Wisconsin
  - Aurora Cardiovascular Services, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects are consented and randomized before the pacing prodecure. They may have been excluded (considered screen fails) if they end up not having the procedure or being identified as inappropriate once the procedure began. 50 Consented and 41 Randomized.
Groups:
- Dual Site LV Pacing First, Then BiV Pacing, Then Physician Dis: Prospective randomized blinded crossover study of patients meeting current CRT-D indication implanted with Dual LV pacing leads compared to BiV pacing.
  Randomized to Dual Site LV Pacing for three months then crossed over to standard BIV pacing for three months then programmed per physician discretion for the remainder three months.
- BiV Pacing First, Then Dual Site LV Pacing, Then Physician Dis: Prospective randomized blinded crossover study of patients meeting current CRT-D indication implanted with Dual LV pacing leads compared to BiV pacing.
  Randomized to standard BiV pacing for three months then crossed over to Dual LV pacing for three months, then programmed per physician discretion for the remainder of the study.
Period: Baseline to 3 Months
Arm/Group | Dual Site LV Pacing First, Then BiV Pacing, Then Physician Dis | BiV Pacing First, Then Dual Site LV Pacing, Then Physician Dis
Started | 19 | 22
Completed | 19 | 22
Not Completed | 0 | 0
Period: 3 to 6 Months
Arm/Group | Dual Site LV Pacing First, Then BiV Pacing, Then Physician Dis | BiV Pacing First, Then Dual Site LV Pacing, Then Physician Dis
Started | 19 | 22
Completed | 19 | 20
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2
Period: 6 Months to Study Completion
Arm/Group | Dual Site LV Pacing First, Then BiV Pacing, Then Physician Dis | BiV Pacing First, Then Dual Site LV Pacing, Then Physician Dis
Started | 19 | 20
Completed | 19 | 18
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Population: Includes both randomized groups, Group A: Randomized to Dual LV pacing for three months then crossed over to Standard BiV pacing for three months, then programmed at the physician discretion. Group B: Randomized to Standard BiV pacing for three months then crossed over to Dual LV pacing for three months, then programmed to physician discretion.
Groups:
- All Study Participants: Prospective randomized blinded crossover study of patients meeting current CRT-D indication implanted with Dual LV pacing leads compared to BiV pacing.
  Randomized to Arm A: Dual Site LV Pacing for three months then crossed over to standard BIV pacing for three months then programmed per physician discretion for the remainder three months. Randomized to Arm B: Randomized to standard BiV pacing for three months then crossed over to Dual LV pacing for three months, then programmed per physician discretion for the remainder of the study.
Arm/Group | All Study Participants
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.5 (10.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Left Ventricular End Systolic Volume (LVESV)
Description: The change in LVESV during the single and dual site LV pacing phases from baseline will be compared. The baseline for the second phase of the cross-over will be the end of phase one rather than the baseline done at time of randomization. Thus, the study will compare the incremental (or decremental) benefit of the alternate LV pacing configuration in each patient.
Time Frame: At 6 months to one year
Population: Analysis population was based on the two randomized groups per the protocol.
Measure: Mean (Standard Deviation); unit: ml
Arm/Group | Dual Site LV Pacing | BiV Pacing
Number analyzed (Participants) | 17 | 14
ml | -28.16 (14.62) | -25.91 (27.84)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse Events were collected per intervention.
Groups:
- Dual Site LV Pacing: Prospective randomized blinded crossover study of patients meeting current CRT-D indication implanted with Dual LV pacing leads compared to BiV pacing.
  Randomized to Dual Site LV Pacing for three months then crossed over to standard BIV pacing for three months then programmed per physician discretion for the remainder three months.
- BiV Pacing: Prospective randomized blinded crossover study of patients meeting current CRT-D indication implanted with Dual LV pacing leads compared to BiV pacing.
  Randomized to standard BiV pacing for three months then crossed over to Dual LV pacing for three months, then programmed per physician discretion for the remainder of the study.
Arm/Group | Dual Site LV Pacing | BiV Pacing
Serious Adverse Events (participants affected / at risk) | 3/41 | 3/41
Other Adverse Events (participants affected / at risk) | 10/41 | 3/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dual Site LV Pacing (N=41) | BiV Pacing (N=41)
Syncope (Vascular disorders) | 0 (0) | 1 (1) — A disorder characterized by spontaneous loss of consciousness caused by insufficient blood supply to the brain.
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) — disorder characterized by an uncomfortable sensation of difficulty breathing.
Heart failure (Cardiac disorders) | 2 (2) | 0 (0) — (exacerbation of existing condition) A disorder characterized by the inability of the heart to pump blood at an adequate volume to meet tissue metabolic requirements, or, the ability to do so only at an elevation in the filling pressure.
Death (General disorders) | 1 (1) | 0 (0) — (not related to investigation)
Multi-organ failure (General disorders) | 1 (1) | 0 (0) — (not related to investigation) A disorder characterized by progressive deterioration of the lungs, liver, kidney and clotting mechanisms.
Sepsis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — A disorder characterized by the presence of pathogenic microorganisms in the blood stream that cause a rapidly progressing systemic reaction that may lead to shock.
Fall (General disorders) | 0 (0) | 2 (2) — A finding of sudden movement downward, usually resulting in injury.
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 2 (2) — A disorder characterized by pathological irregularities in the cardiac conduction system.
Hyperkalemia (Renal and urinary disorders) | 0 (0) | 1 (1) — A disorder characterized by laboratory test results that indicate an elevation in the concentration of potassium in the blood; associated with kidney failure or sometimes with the use of diuretic drugs.
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) — A disorder characterized by the reflexive act of ejecting the contents of the stomach through the mouth.
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) — GI bleed, non specific
Stomach pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — A disorder characterized by a sensation of marked discomfort in the stomach.
Rectal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) — A disorder characterized by an abnormal communication between the rectum and another organ or anatomic site.
ICD shock (Cardiac disorders) | 1 (1) | 1 (1)
Lead dislodgement (Cardiac disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — A disorder characterized by an reduction in the amount of hemoglobin in 100 ml of blood.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dual Site LV Pacing (N=41) | BiV Pacing (N=41)
Diaphragmatic Stimulation (General disorders) | 7 (7) | 3 (3) — Simulation of the phrenic nerve or diaphragm by a pacing output pulse, causing a hiccough-like reaction.
Fatigue (General disorders) | 3 (3) | 0 (0) — A disorder characterized by a state of generalized weakness with a pronounced inability to summon sufficient energy to accomplish daily activities.

LIMITATIONS AND CAVEATS:
Study terminated early form administrative reasons (no safety concerns), no analysis was completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes